CLINICAL TRIAL: NCT05633056
Title: Adaptive Evaluation of mHealth and Conventional Adherence Support Interventions to Optimize Outcome With New Treatment Regimens for Drug-resistant Tuberculosis and HIV in South Africa
Brief Title: An Adaptive Randomized Controlled Trial
Acronym: ADAP-TIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centre for the AIDS Programme of Research in South Africa (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Max O'Donnell, MD,MPH,Principal investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAT8513; CAP262 (Other: University of KwaZulu Natal-Biomedical Research Ethics Committee); 1R01AI167795 (NIH)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Multi Drug Resistant Tuberculosis; HIV Infections
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; HIV Infections

STUDY DESIGN:
Intervention Model Description: An adaptive, randomized controlled trial comparing the effectiveness of 4 adherence support intervention arms. Interventions arms include: enhanced standard of care; psychosocial support; mHealth using cellular-enabled electronic dose monitoring; combined mHealth psychosocial support. Level of support will be adjusted using a differentiated service delivery (DSD)- informed assessment of treatment support needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced standard of care (No Intervention): * Care from trained and supported physicians, nurses, and social workers who have received repeated trainings from study staff on medical and behavioral aspects of DR-TB HIV care, which will be documented in terms of date, attendance, and content
  * All participants who receive care as inpatients will receive an orientation to DR-TB treatment in form of a group session designed to impart key behavioral information and health knowledge about the disease, treatment, and skills to obtain optimal outcome.
  * Discharge counselling session will be conducted prior to discharge.
  * Study participants will complete study assessments at baseline (enrollment) and monthly for the first six months.
- Psychosocial support (Other): * In addition to Arm 1
  * Participants will participate in individual counseling aligned with their monthly clinic visit.
  * Individual counseling will use motivational interviewing (MI) techniques, based on the 4-part engaging, focusing, evoking and planning approach for each participant.
  * Home visits will be conducted (if warranted/consented for by the participant) by the same trained counselors known to patients.
  * Adherence support groups will be facilitated by counselors trained in group facilitation methods; group curriculum will include 6 sessions (monthly, gender specific, structured adherence support groups) that focus on practical topics.
  * Discharge planning (if inpatient)
  * Community treatment planning (if outpatient)
  Interventions: Behavioral: Adherence support intevention
- mHealth (Other): * In addition to Arm 1
  * Participants will receive x 2 portable Wisepill devices. (x1 for MDR-TB treatment and x1 for ART).
  A Wisepill device is an RT2000 cellular-enabled electronic pill boxes using 2G/3G cellular network.
  * Participants will select a text message reminder from a guided menu of choices and receive a weekly text message encouraging adherence.
  * Participants will receive a study call to support regular adherence. Participants will be assessed weekly. Less than 85% observed/expected doses will be considered at risk for non-adherence and the intervention will be increased.
  Interventions: Behavioral: Adherence support intevention
- mHealth and Psychosocial support (Other): Combination of Arm 2 and Arm 3.
  Interventions: Behavioral: Adherence support intevention

INTERVENTIONS:
Behavioral: Adherence support intevention — Compare the effects of adherence support interventions on clinical and biological endpoints using an adaptive randomized platform.
  Arms: Psychosocial support; mHealth; mHealth and Psychosocial support

SUMMARY:
This is a prospective, adaptive, randomized controlled trial comparing the effectiveness of 4 intervention arms on a combined endpoint in adults with confirmed MDR-TB HIV initiating Bedaquiline-containing MDR-TB treatment regimens and on ART (integrase strand transfer inhibitor (INSTI)-based fixed dose combination therapy) in KwaZulu-Natal, South Africa. Interventions arms include: enhanced standard of care; psychosocial support; mHealth using cellular-enabled electronic dose monitoring; combined mHealth psychosocial support. Level of support will be adjusted using a differentiated service delivery (DSD)- informed assessment of treatment support needs.

DETAILED DESCRIPTION:
This study will follow a 4-arm Bayesian, adaptive trial design. As patients are enrolled, they will be randomized into one of the four arms.

The study will be carried out within a common structure to allow for efficient enrollment and analysis. The overall structure is a 4-arm adaptive platform of mHealth and psychosocial adherence support interventions informed by a differentiated service delivery (DSD) approach.

Aim 1 is an adaptive study of mHealth and psychosocial adherence support interventions using a Bayesian adaptive design to allow comparison of elements of the intervention separately and in combination. Aim 1 participants will be randomized into one of 4 arms and followed monthly through the 6 months of intervention, then through the end of treatment telephonically, with an additional in-person visit to establish the primary outcome. Primary outcome is a combined clinical/biological outcome at 12 months described below. Hypothesis 1a utilizes all participants while 1b utilizes only those in the mHealth intervention arms (3+4) since granular EDM-measured adherence is required.

ELIGIBILITY:
Inclusion Criteria:

1. Culture or molecular test positive for MTB
2. Molecular test positive for HIV or a documented HIV positive history
3. Drug-susceptibility testing by molecular (i.e. GeneXpert MTB/RIF) or conventional testing consistent with at least rifampicin-resistant TB,
4. Initiating treatment with a Bedaquiline -containing TB regimen within 4 weeks of enrollment and first-time being treated with BDQ
5. On treatment with Antiretroviral Therapy (ART) regimen, including dolutegravir-containing combination Antiretroviral Therapy regimen (i.e. Tenofovir-Lamivudine-Dolutergravir), or starting within 4 weeks of enrollment,
6. Capacity for informed consent in either isiZulu or English

Exclusion Criteria:

1. Pregnancy
2. Prisoners
3. Discretion of IOR or clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Biological outcome | 06 months
  TB culture conversion
Clinical outcome | 12 months
  Survival
Biological outcome | 12 months
  HIV viral load
Clinical outcome | 12 months
  Retention in care
Biological outcome | 12 months
  TB culture conversion

CONTACTS AND LOCATIONS:
Overall Officials: Max O'Donnell, Prof, Principal Investigator — University of Columbia
Locations (1):
- King DinuZulu Hospital, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diacon AH, Pym A, Grobusch MP, de los Rios JM, Gotuzzo E, Vasilyeva I, Leimane V, Andries K, Bakare N, De Marez T, Haxaire-Theeuwes M, Lounis N, Meyvisch P, De Paepe E, van Heeswijk RP, Dannemann B; TMC207-C208 Study Group. Multidrug-resistant tuberculosis and culture conversion with bedaquiline. N Engl J Med. 2014 Aug 21;371(8):723-32. doi: 10.1056/NEJMoa1313865. PMID 25140958
- [Background] O'Donnell MR, Padayatchi N, Daftary A, Orrell C, Dooley KE, Rivet Amico K, Friedland G. Antiretroviral switching and bedaquiline treatment of drug-resistant tuberculosis HIV co-infection. Lancet HIV. 2019 Mar;6(3):e201-e204. doi: 10.1016/S2352-3018(19)30035-9. PMID 30846058
- [Background] Calmy A, Tovar Sanchez T, Kouanfack C, Mpoudi-Etame M, Leroy S, Perrineau S, Lantche Wandji M, Tetsa Tata D, Omgba Bassega P, Abong Bwenda T, Varloteaux M, Tongo M, Mpoudi-Ngole E, Montoyo A, Mercier N, LeMoing V, Peeters M, Reynes J, Delaporte E; New Antiretroviral and Monitoring Strategies in HIV-infected Adults in Low-Income Countries (NAMSAL) ANRS 12313 Study Group. Dolutegravir-based and low-dose efavirenz-based regimen for the initial treatment of HIV-1 infection (NAMSAL): week 96 results from a two-group, multicentre, randomised, open label, phase 3 non-inferiority trial in Cameroon. Lancet HIV. 2020 Oct;7(10):e677-e687. doi: 10.1016/S2352-3018(20)30238-1. PMID 33010241
- [Background] NAMSAL ANRS 12313 Study Group; Kouanfack C, Mpoudi-Etame M, Omgba Bassega P, Eymard-Duvernay S, Leroy S, Boyer S, Peeters M, Calmy A, Delaporte E. Dolutegravir-Based or Low-Dose Efavirenz-Based Regimen for the Treatment of HIV-1. N Engl J Med. 2019 Aug 29;381(9):816-826. doi: 10.1056/NEJMoa1904340. Epub 2019 Jul 24. PMID 31339676
- [Background] Nimmo C, Millard J, Brien K, Moodley S, van Dorp L, Lutchminarain K, Wolf A, Grant AD, Balloux F, Pym AS, Padayatchi N, O'Donnell M. Bedaquiline resistance in drug-resistant tuberculosis HIV co-infected patients. Eur Respir J. 2020 Jun 4;55(6):1902383. doi: 10.1183/13993003.02383-2019. Print 2020 Jun. PMID 32060065
- [Background] Nimmo C, Millard J, van Dorp L, Brien K, Moodley S, Wolf A, Grant AD, Padayatchi N, Pym AS, Balloux F, O'Donnell M. Population-level emergence of bedaquiline and clofazimine resistance-associated variants among patients with drug-resistant tuberculosis in southern Africa: a phenotypic and phylogenetic analysis. Lancet Microbe. 2020 Aug;1(4):e165-e174. doi: 10.1016/S2666-5247(20)30031-8. PMID 32803174
- [Background] WHO. World Health Organization. Global tuberculosis report 2020. 2020.
- [Background] Saunders MJ, Evans CA. COVID-19, tuberculosis and poverty: preventing a perfect storm. Eur Respir J. 2020 Jul 9;56(1):2001348. doi: 10.1183/13993003.01348-2020. Print 2020 Jul. PMID 32444399
- [Background] Gupta RK, Lucas SB, Fielding KL, Lawn SD. Prevalence of tuberculosis in post-mortem studies of HIV-infected adults and children in resource-limited settings: a systematic review and meta-analysis. AIDS. 2015 Sep 24;29(15):1987-2002. doi: 10.1097/QAD.0000000000000802. PMID 26266773
- [Background] Zellweger JP, Heinzer R, Touray M, Vidondo B, Altpeter E. Intra-observer and overall agreement in the radiological assessment of tuberculosis. Int J Tuberc Lung Dis. 2006 Oct;10(10):1123-6. PMID 17044205
- [Background] Mabhula A, Singh V. Drug-resistance in Mycobacterium tuberculosis: where we stand. Medchemcomm. 2019 Jun 11;10(8):1342-1360. doi: 10.1039/c9md00057g. eCollection 2019 Aug 1. PMID 31534654
- [Background] Ahuja SD, Ashkin D, Avendano M, Banerjee R, Bauer M, Bayona JN, Becerra MC, Benedetti A, Burgos M, Centis R, Chan ED, Chiang CY, Cox H, D'Ambrosio L, DeRiemer K, Dung NH, Enarson D, Falzon D, Flanagan K, Flood J, Garcia-Garcia ML, Gandhi N, Granich RM, Hollm-Delgado MG, Holtz TH, Iseman MD, Jarlsberg LG, Keshavjee S, Kim HR, Koh WJ, Lancaster J, Lange C, de Lange WC, Leimane V, Leung CC, Li J, Menzies D, Migliori GB, Mishustin SP, Mitnick CD, Narita M, O'Riordan P, Pai M, Palmero D, Park SK, Pasvol G, Pena J, Perez-Guzman C, Quelapio MI, Ponce-de-Leon A, Riekstina V, Robert J, Royce S, Schaaf HS, Seung KJ, Shah L, Shim TS, Shin SS, Shiraishi Y, Sifuentes-Osornio J, Sotgiu G, Strand MJ, Tabarsi P, Tupasi TE, van Altena R, Van der Walt M, Van der Werf TS, Vargas MH, Viiklepp P, Westenhouse J, Yew WW, Yim JJ; Collaborative Group for Meta-Analysis of Individual Patient Data in MDR-TB. Multidrug resistant pulmonary tuberculosis treatment regimens and patient outcomes: an individual patient data meta-analysis of 9,153 patients. PLoS Med. 2012;9(8):e1001300. doi: 10.1371/journal.pmed.1001300. Epub 2012 Aug 28. PMID 22952439
- [Background] Cohen T, Murray M, Wallengren K, Alvarez GG, Samuel EY, Wilson D. The prevalence and drug sensitivity of tuberculosis among patients dying in hospital in KwaZulu-Natal, South Africa: a postmortem study. PLoS Med. 2010 Jun 22;7(6):e1000296. doi: 10.1371/journal.pmed.1000296. PMID 20582324
- [Background] Abdool Karim Q, Abdool Karim SS. COVID-19 affects HIV and tuberculosis care. Science. 2020 Jul 24;369(6502):366-368. doi: 10.1126/science.abd1072. No abstract available. PMID 32703860
- [Background] Basu S, Andrews JR, Poolman EM, Gandhi NR, Shah NS, Moll A, Moodley P, Galvani AP, Friedland GH. Prevention of nosocomial transmission of extensively drug-resistant tuberculosis in rural South African district hospitals: an epidemiological modelling study. Lancet. 2007 Oct 27;370(9597):1500-7. doi: 10.1016/S0140-6736(07)61636-5. PMID 17964351
- [Background] Shah NS, Auld SC, Brust JC, Mathema B, Ismail N, Moodley P, Mlisana K, Allana S, Campbell A, Mthiyane T, Morris N, Mpangase P, van der Meulen H, Omar SV, Brown TS, Narechania A, Shaskina E, Kapwata T, Kreiswirth B, Gandhi NR. Transmission of Extensively Drug-Resistant Tuberculosis in South Africa. N Engl J Med. 2017 Jan 19;376(3):243-253. doi: 10.1056/NEJMoa1604544. PMID 28099825
- [Background] Adane AA, Alene KA, Koye DN, Zeleke BM. Non-adherence to anti-tuberculosis treatment and determinant factors among patients with tuberculosis in northwest Ethiopia. PLoS One. 2013 Nov 11;8(11):e78791. doi: 10.1371/journal.pone.0078791. eCollection 2013. PMID 24244364
- [Background] Kulkarni P, Akarte S, Mankeshwar R, Bhawalkar J, Banerjee A, Kulkarni A. Non-adherence of new pulmonary tuberculosis patients to anti-tuberculosis treatment. Ann Med Health Sci Res. 2013 Jan;3(1):67-74. doi: 10.4103/2141-9248.109507. PMID 23634333
- [Background] Gandhi NR, Moll A, Sturm AW, Pawinski R, Govender T, Lalloo U, Zeller K, Andrews J, Friedland G. Extensively drug-resistant tuberculosis as a cause of death in patients co-infected with tuberculosis and HIV in a rural area of South Africa. Lancet. 2006 Nov 4;368(9547):1575-80. doi: 10.1016/S0140-6736(06)69573-1. PMID 17084757
- [Background] Gardner EM, McLees MP, Steiner JF, Del Rio C, Burman WJ. The spectrum of engagement in HIV care and its relevance to test-and-treat strategies for prevention of HIV infection. Clin Infect Dis. 2011 Mar 15;52(6):793-800. doi: 10.1093/cid/ciq243. PMID 21367734
- [Background] Senthilingam M, Pietersen E, McNerney R, Te Riele J, Sedres P, Wilson R, Dheda K. Lifestyle, attitudes and needs of uncured XDR-TB patients living in the communities of South Africa: a qualitative study. Trop Med Int Health. 2015 Sep;20(9):1155-1161. doi: 10.1111/tmi.12532. Epub 2015 May 18. PMID 25941041
- [Background] Daftary A, Padayatchi N, O'Donnell M. Preferential adherence to antiretroviral therapy over tuberculosis treatment: a qualitative study of drug-resistant TB/HIV co-infected patients in South Africa. Glob Public Health. 2014;9(9):1107-16. doi: 10.1080/17441692.2014.934266. Epub 2014 Jul 18. PMID 25035943
- [Background] Daftary A, Padayatchi N. Social constraints to TB/HIV healthcare: accounts from coinfected patients in South Africa. AIDS Care. 2012;24(12):1480-6. doi: 10.1080/09540121.2012.672719. Epub 2012 Apr 24. PMID 22530855
- [Background] Mansoor LE, Karim QA, Werner L, Madlala B, Ngcobo N, Cornman DH, Amico KR, Fisher J, Fisher WA, Macqueen KM, Karim SS. Impact of an adherence intervention on the effectiveness of tenofovir gel in the CAPRISA 004 trial. AIDS Behav. 2014 May;18(5):841-8. doi: 10.1007/s10461-014-0752-9. PMID 24633717
- [Background] O'Laughlin KN, Wyatt MA, Kaaya S, Bangsberg DR, Ware NC. How treatment partners help: social analysis of an African adherence support intervention. AIDS Behav. 2012 Jul;16(5):1308-15. doi: 10.1007/s10461-011-0038-4. PMID 21947835
- [Background] Brust JC, Gandhi NR, Carrara H, Osburn G, Padayatchi N. High treatment failure and default rates for patients with multidrug-resistant tuberculosis in KwaZulu-Natal, South Africa, 2000-2003. Int J Tuberc Lung Dis. 2010 Apr;14(4):413-9. PMID 20202298
- [Background] Nelson KN, Shah NS, Mathema B, Ismail N, Brust JCM, Brown TS, Auld SC, Omar SV, Morris N, Campbell A, Allana S, Moodley P, Mlisana K, Gandhi NR. Spatial Patterns of Extensively Drug-Resistant Tuberculosis Transmission in KwaZulu-Natal, South Africa. J Infect Dis. 2018 Nov 5;218(12):1964-1973. doi: 10.1093/infdis/jiy394. PMID 29961879
- [Background] Brown TS, Challagundla L, Baugh EH, Omar SV, Mustaev A, Auld SC, Shah NS, Kreiswirth BN, Brust JCM, Nelson KN, Narechania A, Kurepina N, Mlisana K, Bonneau R, Eldholm V, Ismail N, Kolokotronis SO, Robinson DA, Gandhi NR, Mathema B. Pre-detection history of extensively drug-resistant tuberculosis in KwaZulu-Natal, South Africa. Proc Natl Acad Sci U S A. 2019 Nov 12;116(46):23284-23291. doi: 10.1073/pnas.1906636116. Epub 2019 Oct 28. PMID 31659018
- [Background] Isaakidis P, Casas EC, Das M, Tseretopoulou X, Ntzani EE, Ford N. Treatment outcomes for HIV and MDR-TB co-infected adults and children: systematic review and meta-analysis. Int J Tuberc Lung Dis. 2015 Aug;19(8):969-78. doi: 10.5588/ijtld.15.0123. PMID 26162364
- [Background] Singh A, Prasad R, Balasubramanian V, Gupta N. Drug-Resistant Tuberculosis and HIV Infection: Current Perspectives. HIV AIDS (Auckl). 2020 Jan 13;12:9-31. doi: 10.2147/HIV.S193059. eCollection 2020. PMID 32021483
- [Background] Walmsley SL, Antela A, Clumeck N, Duiculescu D, Eberhard A, Gutierrez F, Hocqueloux L, Maggiolo F, Sandkovsky U, Granier C, Pappa K, Wynne B, Min S, Nichols G; SINGLE Investigators. Dolutegravir plus abacavir-lamivudine for the treatment of HIV-1 infection. N Engl J Med. 2013 Nov 7;369(19):1807-18. doi: 10.1056/NEJMoa1215541. PMID 24195548
- [Background] Vitoria M, Hill A, Ford N, Doherty M, Clayden P, Venter F, Ripin D, Flexner C, Domanico PL. The transition to dolutegravir and other new antiretrovirals in low-income and middle-income countries: what are the issues? AIDS. 2018 Jul 31;32(12):1551-1561. doi: 10.1097/QAD.0000000000001845. PMID 29746295
- [Background] Schnippel K, Ndjeka N, Maartens G, Meintjes G, Master I, Ismail N, Hughes J, Ferreira H, Padanilam X, Romero R, Te Riele J, Conradie F. Effect of bedaquiline on mortality in South African patients with drug-resistant tuberculosis: a retrospective cohort study. Lancet Respir Med. 2018 Sep;6(9):699-706. doi: 10.1016/S2213-2600(18)30235-2. Epub 2018 Jul 11. PMID 30001994
- [Background] Meireles MV, Pascom ARP, Duarte EC, McFarland W. Comparative effectiveness of first-line antiretroviral therapy: results from a large real-world cohort after the implementation of dolutegravir. AIDS. 2019 Aug 1;33(10):1663-1668. doi: 10.1097/QAD.0000000000002254. PMID 31082860
- [Background] Howell EM, Kigozi NG, Heunis JC. Community-based directly observed treatment for TB patients to improve HIV services: a cross-sectional study in a South African province. BMC Health Serv Res. 2018 Apr 7;18(1):255. doi: 10.1186/s12913-018-3074-1. PMID 29625569
- [Background] Mannheimer S, Friedland G, Matts J, Child C, Chesney M. The consistency of adherence to antiretroviral therapy predicts biologic outcomes for human immunodeficiency virus-infected persons in clinical trials. Clin Infect Dis. 2002 Apr 15;34(8):1115-21. doi: 10.1086/339074. Epub 2002 Mar 11. PMID 11915001
- [Background] Alipanah N, Jarlsberg L, Miller C, Linh NN, Falzon D, Jaramillo E, Nahid P. Adherence interventions and outcomes of tuberculosis treatment: A systematic review and meta-analysis of trials and observational studies. PLoS Med. 2018 Jul 3;15(7):e1002595. doi: 10.1371/journal.pmed.1002595. eCollection 2018 Jul. PMID 29969463
- [Background] Iacob SA, Iacob DG, Jugulete G. Improving the Adherence to Antiretroviral Therapy, a Difficult but Essential Task for a Successful HIV Treatment-Clinical Points of View and Practical Considerations. Front Pharmacol. 2017 Nov 23;8:831. doi: 10.3389/fphar.2017.00831. eCollection 2017. PMID 29218008
- [Background] van den Boogaard J, Boeree MJ, Kibiki GS, Aarnoutse RE. The complexity of the adherence-response relationship in tuberculosis treatment: why are we still in the dark and how can we get out? Trop Med Int Health. 2011 Jun;16(6):693-8. doi: 10.1111/j.1365-3156.2011.02755.x. Epub 2011 Mar 6. PMID 21375681
- [Background] O'Donnell MR, Daftary A, Frick M, Hirsch-Moverman Y, Amico KR, Senthilingam M, Wolf A, Metcalfe JZ, Isaakidis P, Davis JL, Zelnick JR, Brust JC, Naidu N, Garretson M, Bangsberg DR, Padayatchi N, Friedland G. Re-inventing adherence: toward a patient-centered model of care for drug-resistant tuberculosis and HIV. Int J Tuberc Lung Dis. 2016 Apr;20(4):430-4. doi: 10.5588/ijtld.15.0360. PMID 26970149
- [Background] Stephens F, Gandhi NR, Brust JCM, Mlisana K, Moodley P, Allana S, Campbell A, Shah S. Treatment Adherence Among Persons Receiving Concurrent Multidrug-Resistant Tuberculosis and HIV Treatment in KwaZulu-Natal, South Africa. J Acquir Immune Defic Syndr. 2019 Oct 1;82(2):124-130. doi: 10.1097/QAI.0000000000002120. PMID 31513073
- [Background] O'Donnell MR, Wolf A, Werner L, Horsburgh CR, Padayatchi N. Adherence in the treatment of patients with extensively drug-resistant tuberculosis and HIV in South Africa: a prospective cohort study. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):22-9. doi: 10.1097/QAI.0000000000000221. PMID 24872138
- [Background] Daftary A, Mondal S, Zelnick J, Friedland G, Seepamore B, Boodhram R, Amico KR, Padayatchi N, O'Donnell MR. Dynamic needs and challenges of people with drug-resistant tuberculosis and HIV in South Africa: a qualitative study. Lancet Glob Health. 2021 Apr;9(4):e479-e488. doi: 10.1016/S2214-109X(20)30548-9. PMID 33740409
- [Background] Law S, Daftary A, O'Donnell M, Padayatchi N, Calzavara L, Menzies D. Interventions to improve retention-in-care and treatment adherence among patients with drug-resistant tuberculosis: a systematic review. Eur Respir J. 2019 Jan 10;53(1):1801030. doi: 10.1183/13993003.01030-2018. Print 2019 Jan. PMID 30309972
- [Background] Bionghi N, Daftary A, Maharaj B, Msibi Z, Amico KR, Friedland G, Orrell C, Padayatchi N, O'Donnell MR. Pilot evaluation of a second-generation electronic pill box for adherence to Bedaquiline and antiretroviral therapy in drug-resistant TB/HIV co-infected patients in KwaZulu-Natal, South Africa. BMC Infect Dis. 2018 Apr 11;18(1):171. doi: 10.1186/s12879-018-3080-2. PMID 29642874
- [Background] MacCarthy S, Mendoza-Graf A, Saya U, Samba C, Birungi J, Okoboi S, Linnemayr S. Lessons learned from a mobile technology-based intervention informed by behavioral economics to improve ART adherence among youth in Uganda. AIDS Care. 2020 May;32(5):616-622. doi: 10.1080/09540121.2019.1622630. Epub 2019 May 28. PMID 31137959
- [Background] Haberer JE, Sabin L, Amico KR, Orrell C, Galarraga O, Tsai AC, Vreeman RC, Wilson I, Sam-Agudu NA, Blaschke TF, Vrijens B, Mellins CA, Remien RH, Weiser SD, Lowenthal E, Stirratt MJ, Sow PS, Thomas B, Ford N, Mills E, Lester R, Nachega JB, Bwana BM, Ssewamala F, Mbuagbaw L, Munderi P, Geng E, Bangsberg DR. Improving antiretroviral therapy adherence in resource-limited settings at scale: a discussion of interventions and recommendations. J Int AIDS Soc. 2017 Mar 22;20(1):21371. doi: 10.7448/IAS.20.1.21371. eCollection 2017. PMID 28630651
- [Background] Shaw S, Amico KR. Antiretroviral Therapy Adherence Enhancing Interventions for Adolescents and Young Adults 13-24 Years of Age: A Review of the Evidence Base. J Acquir Immune Defic Syndr. 2016 Aug 1;72(4):387-99. doi: 10.1097/QAI.0000000000000977. PMID 26959190
- [Background] Cooper V, Clatworthy J, Whetham J, Consortium E. mHealth Interventions To Support Self-Management In HIV: A Systematic Review. Open AIDS J. 2017 Nov 21;11:119-132. doi: 10.2174/1874613601711010119. eCollection 2017. PMID 29290888
- [Background] Chiang N, Guo M, Amico KR, Atkins L, Lester RT. Interactive Two-Way mHealth Interventions for Improving Medication Adherence: An Evaluation Using The Behaviour Change Wheel Framework. JMIR Mhealth Uhealth. 2018 Apr 12;6(4):e87. doi: 10.2196/mhealth.9187. PMID 29650504
- [Background] Haldane V, Koh JJK, Srivastava A, Teo KWQ, Tan YG, Cheng RX, Yap YC, Ong PS, Van Dam RM, Foo JM, Muller-Riemenschneider F, Koh GC, Foong PS, Perel P, Legido-Quigley H. User Preferences and Persona Design for an mHealth Intervention to Support Adherence to Cardiovascular Disease Medication in Singapore: A Multi-Method Study. JMIR Mhealth Uhealth. 2019 May 28;7(5):e10465. doi: 10.2196/10465. PMID 31140445
- [Background] Brewer LC, Jenkins S, Lackore K, Johnson J, Jones C, Cooper LA, Radecki Breitkopf C, Hayes SN, Patten C. mHealth Intervention Promoting Cardiovascular Health Among African-Americans: Recruitment and Baseline Characteristics of a Pilot Study. JMIR Res Protoc. 2018 Jan 31;7(1):e31. doi: 10.2196/resprot.8842. PMID 29386174
- [Background] Zhuang Q, Chen F, Wang T. Effectiveness of short message service intervention to improve glycated hemoglobin control and medication adherence in type-2 diabetes: A meta-analysis of prospective studies. Prim Care Diabetes. 2020 Aug;14(4):356-363. doi: 10.1016/j.pcd.2019.09.007. Epub 2019 Oct 23. PMID 31653588
- [Background] Menon V, Selvakumar N, Kattimani S, Andrade C. Therapeutic effects of mobile-based text message reminders for medication adherence in bipolar I disorder: Are they maintained after intervention cessation? J Psychiatr Res. 2018 Sep;104:163-168. doi: 10.1016/j.jpsychires.2018.07.013. Epub 2018 Jul 26. PMID 30081390
- [Background] Xiao Q, Wang J, Chiang V, Choi T, Wang Y, Sun L, Wu Y. Effectiveness of mHealth Interventions for Asthma Self-Management: A Systematic Review and Meta-Analysis. Stud Health Technol Inform. 2018;250:144-145. PMID 29857410
- [Background] Schindler-Ruwisch JM, Roess A, Robert RC, Napolitano MA, Chiang S. Social Support for Breastfeeding in the Era of mHealth: A Content Analysis. J Hum Lact. 2018 Aug;34(3):543-555. doi: 10.1177/0890334418773302. Epub 2018 May 22. PMID 29787686
- [Background] Zelnick JR, Seepamore B, Daftary A, Amico KR, Bhengu X, Friedland G, Padayatchi N, Naidoo K, O'Donnell MR. Training social workers to enhance patient-centered care for drug-resistant TB-HIV in South Africa. Public Health Action. 2018 Mar 21;8(1):25-27. doi: 10.5588/pha.17.0114. PMID 29581940
- [Background] Rabkin M, Howard AA, Ehrenkranz P, Fernandez LG, Preko P, Singh V, Tomlinson HL, El-Sadr WM. Leveraging differentiated HIV service delivery to expand tuberculosis preventive treatment: a call to action. Int J Tuberc Lung Dis. 2020 Feb 1;24(2):165-169. doi: 10.5588/ijtld.19.0595. PMID 32127099
- [Background] Ehrenkranz P, Grimsrud A, Holmes CB, Preko P, Rabkin M. Expanding the Vision for Differentiated Service Delivery: A Call for More Inclusive and Truly Patient-Centered Care for People Living With HIV. J Acquir Immune Defic Syndr. 2021 Feb 1;86(2):147-152. doi: 10.1097/QAI.0000000000002549. PMID 33136818
- [Background] Ehrenkranz P, Grimsrud A, Rabkin M. Differentiated service delivery: navigating the path to scale. Curr Opin HIV AIDS. 2019 Jan;14(1):60-65. doi: 10.1097/COH.0000000000000509. PMID 30394947
- [Background] Roy M, Bolton Moore C, Sikazwe I, Holmes CB. A Review of Differentiated Service Delivery for HIV Treatment: Effectiveness, Mechanisms, Targeting, and Scale. Curr HIV/AIDS Rep. 2019 Aug;16(4):324-334. doi: 10.1007/s11904-019-00454-5. PMID 31230342
- [Background] E. G. Stigma: notes on the management of spoiled identity. USA: Simons & Schuster, Inc.; 1963
- [Background] Pescosolido BA, Martin JK. The Stigma Complex. Annu Rev Sociol. 2015 Aug;41:87-116. doi: 10.1146/annurev-soc-071312-145702. Epub 2015 May 4. PMID 26855471
- [Background] Parker R, Aggleton P. HIV and AIDS-related stigma and discrimination: a conceptual framework and implications for action. Soc Sci Med. 2003 Jul;57(1):13-24. doi: 10.1016/s0277-9536(02)00304-0. PMID 12753813
- [Background] Stangl AL, Lloyd JK, Brady LM, Holland CE, Baral S. A systematic review of interventions to reduce HIV-related stigma and discrimination from 2002 to 2013: how far have we come? J Int AIDS Soc. 2013 Nov 13;16(3 Suppl 2):18734. doi: 10.7448/IAS.16.3.18734. PMID 24242268
- [Background] Hirsch-Moverman Y, Daftary A, Yuengling KA, Saito S, Ntoane M, Frederix K, Maama LB, Howard AA. Using mHealth for HIV/TB Treatment Support in Lesotho: Enhancing Patient-Provider Communication in the START Study. J Acquir Immune Defic Syndr. 2017 Jan 1;74 Suppl 1(Suppl 1):S37-S43. doi: 10.1097/QAI.0000000000001202. PMID 27930610
- [Background] Edginton ME, Sekatane CS, Goldstein SJ. Patients' beliefs: do they affect tuberculosis control? A study in a rural district of South Africa. Int J Tuberc Lung Dis. 2002 Dec;6(12):1075-82. PMID 12546115
- [Background] Daftary A. HIV and tuberculosis: the construction and management of double stigma. Soc Sci Med. 2012 May;74(10):1512-9. doi: 10.1016/j.socscimed.2012.01.027. Epub 2012 Mar 7. PMID 22444460
- [Background] Nyblade LC. Measuring HIV stigma: existing knowledge and gaps. Psychol Health Med. 2006 Aug;11(3):335-45. doi: 10.1080/13548500600595178. PMID 17130069
- [Background] Gao J, Su PF, Hu F, Cheung SH. Adaptive treatment allocation for comparative clinical studies with recurrent events data. Biometrics. 2020 Mar;76(1):183-196. doi: 10.1111/biom.13117. Epub 2019 Sep 12. PMID 31282997
- [Background] Mansoor LE, Abdool Karim Q, Mngadi KT, Dlamini S, Montague C, Nkomonde N, Mvandaba N, Baxter C, Gengiah TN, Samsunder N, Dawood H, Grobler A, Frohlich JA, Abdool Karim SS. Assessing the implementation effectiveness and safety of 1% tenofovir gel provision through family planning services in KwaZulu-Natal, South Africa: study protocol for an open-label randomized controlled trial. Trials. 2014 Dec 19;15:496. doi: 10.1186/1745-6215-15-496. PMID 25527071
- [Background] Lassi ZS, Kumar R, Mansoor T, Salam RA, Das JK, Bhutta ZA. Essential interventions: implementation strategies and proposed packages of care. Reprod Health. 2014;11 Suppl 1(Suppl 1):S5. doi: 10.1186/1742-4755-11-S1-S5. Epub 2014 Aug 21. PMID 25178110
- [Background] Cheung YK, Inoue LY, Wathen JK, Thall PF. Continuous Bayesian adaptive randomization based on event times with covariates. Stat Med. 2006 Jan 15;25(1):55-70. doi: 10.1002/sim.2247. PMID 16025549
- [Background] Cheung YK, Thall PF. Monitoring the rates of composite events with censored data in phase II clinical trials. Biometrics. 2002 Mar;58(1):89-97. doi: 10.1111/j.0006-341x.2002.00089.x. PMID 11890331
- [Background] Miller WR, Moyers TB. Motivational interviewing and the clinical science of Carl Rogers. J Consult Clin Psychol. 2017 Aug;85(8):757-766. doi: 10.1037/ccp0000179. PMID 28726479
- [Background] Yuengling KA, Padayatchi N, Wolf A, Mathema B, Brown T, Horsburgh CR, O'Donnell MR. Effect of Antiretroviral Therapy on Treatment Outcomes in a Prospective Study of Extensively Drug-Resistant Tuberculosis (XDR-TB) HIV Coinfection Treatment in KwaZulu-Natal, South Africa. J Acquir Immune Defic Syndr. 2018 Dec 1;79(4):474-480. doi: 10.1097/QAI.0000000000001833. PMID 30212394
- [Background] Visser M, Mundell J, de Villiers A, Sikkema K, Jeffery B. Development of structured support groups for HIV-positive women in South Africa. SAHARA J. 2005 Nov;2(3):333-43. doi: 10.1080/17290376.2005.9724858. PMID 17600975
- [Background] Lennon-Dearing R. The Benefits of Women-Only HIV Support Groups. Journal of HIV/AIDS & Social Services. 2008;7(1):27-45
- [Background] THOMPSON WR. ON THE LIKELIHOOD THAT ONE UNKNOWN PROBABILITY EXCEEDS ANOTHER IN VIEW OF THE EVIDENCE OF TWO SAMPLES. Biometrika. 1933;25(3-4):285-94.
- [Background] Moller V, Erstad I. Stigma asociated with tuberculosis in a time of HIV/AIDS: narratives from the Eastern Cape, South Africa. South African Review of Sociology. 2007;38(2):103-19.
- [Background] Companion Handbook to the WHO Guidelines for the Programmatic Management of Drug-Resistant Tuberculosis. Geneva: World Health Organization; 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK247420/ PMID 25320836
- [Background] NIAID Research Agenda Multidrug-Resistant and Extensively Drug-Resistant Tuberculosis. NIAID. 2007.
- [Result] Zelnick JR, Daftary A, Hwang C, Labar AS, Boodhram R, Maharaj B, Wolf AK, Mondal S, Amico KR, Orrell C, Seepamore B, Friedland G, Padayatchi N, O'Donnell MR. Electronic Dose Monitoring Identifies a High-Risk Subpopulation in the Treatment of Drug-resistant Tuberculosis and Human Immunodeficiency Virus. Clin Infect Dis. 2021 Oct 5;73(7):e1901-e1910. doi: 10.1093/cid/ciaa1557. PMID 33053186
- [Derived] Ross J, Perumal R, Wolf A, Zulu M, Guzman K, Seepamore B, Reis K, Nyilana H, Hlathi S, Narasimmulu R, Cheung YKK, Amico KR, Friedland G, Daftary A, Zelnick JR, Naidoo K, O'Donnell MR. Adaptive evaluation of mHealth and conventional adherence support interventions to optimize outcomes with new treatment regimens for drug-resistant tuberculosis and HIV in South Africa (ADAP-TIV): study protocol for an adaptive randomized controlled trial. Trials. 2023 Dec 1;24(1):776. doi: 10.1186/s13063-023-07520-9. PMID 38037105
- See also: WHO World Health Organization. The end of TB strategy.2015 — https://www.who.int/teams/global-tuberculosis-programme/the-end-tb-strategy

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form: Informed Consent Form-English (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT05633056/Prot_ICF_000.pdf
  • Informed Consent Form: English version (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT05633056/ICF_001.pdf